CLINICAL TRIAL: NCT04917289
Title: Circulating Tumor Cell vs. Radiography as the Evidence of Disease Recurrence in Colorectal Cancer Patients Whose Tumor Underwent R0 Resection
Brief Title: CTC vs Radiography as the Evidence of Recurrence in Colorectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZSCTC3
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Patients in this arm will receive treatment or change current adjuvant therapy immediately after detecting CTC.
  Interventions: Drug: Chemotherapy
- Control Arm (No Intervention): Patients in this arm will keep follow-up after detecting CTC until radiology evidence of recurrence appear.

INTERVENTIONS:
Drug: Chemotherapy — Started chemotherapy or change the current adjuvant therapy
  Arms: Treatment Arm

SUMMARY:
This study enrolled patients who underwent R0 resection of tumor and had elevated tumor biomarkers (CEA, CA19-9). After enroll the study, a CTC test will performed and patients who had positive CTC will be randomly assigned to two groups. The control group will continue follow-up until radiological recurrence appear, the treatment group will start treatment or change the current adjuvant regimen. First endpoint is OS. The secondary endpoint is DFS, adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;

Histologically proven colorectal cancer

All the lesion (s) has been R0 resected

Have elevated tumor biomarker (CEA or CA19-9) in three consecutive tests

More than 1 CTC has been detected (including 1)

ECOG 0-1

Hematology tests suggest that they can tolerate chemotherapy

Written informed consent for participation in the trial

Exclusion Criteria:

* Have any radiological evidence of recurrence

Other previous malignancy within 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 year
  Time from randomization to death

SECONDARY OUTCOMES:
Disease free survival | 3 year
  Disease free time from randomization to death or recurrence
Adverse event | 1 year
  CTCAE adverse event of chemotherapy

IPD SHARING:
Plan to Share IPD: Undecided